CLINICAL TRIAL: NCT02284347
Title: NuVent™ Revision Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Surgical Technologies (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TD-09330
Record Dates: First submitted 2014-10-28; First posted 2014-11-06 (Estimated); Results first posted 2016-08-24 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-07

CONDITIONS: Chronic Rhinosinusitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- NuVent™ (Experimental): Revision patients treated with NuVent™
  Interventions: Device: Electromagnetic Sinus Dilation System (NuVent™)

INTERVENTIONS:
Device: Electromagnetic Sinus Dilation System (NuVent™) — NuVent navigation-guided balloon system may be used to locate and move tissue, bone or cartilaginous tissue obstructing the drainage pathways of the frontal, maxillary, and sphenoid sinuses that is scarred, granulated or previously surgically-altered to facilitate dilation of the sinus ostia.

SUMMARY:
This is a prospective, non-randomized, single-arm study designed to assess the safety and device performance of the NuVent navigation-guided balloon system for use in subjects with scarred, granulated, or previously surgically altered tissue (revision).

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 18 years of age.
2. Subject has chronic rhinosinusitis unresponsive to medical therapy and previous sinus surgery.
3. Subject has sinus surgery planned on at least one of the frontal, sphenoid or maxillary sinus ostia.
4. Subject has scarred, granulated or previously surgically altered tissue for which an image-guided balloon tool may be feasible, in the opinion of the Investigator.
5. Subject is willing and able to comply with protocol requirements.

Exclusion Criteria:

1. Subject is pregnant or breastfeeding.
2. Subject is not healthy enough to undergo endoscopic sinus surgery based on the opinion of the Investigator.
3. Subject has sinonasal tumors.
4. Subject is participating in another investigational device, biologic, or drug study and has not completed the primary endpoint(s) or if there is a potential for clinical interference beyond the primary endpoint.
5. Subject lacks capacity to consent to participation in this research himself/herself.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2014-12; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | NuVent™
Started | 51
Completed | 48
Not Completed | 3
Not completed — Lost to Follow-up | 2
Not completed — Withdrawn prior to treatment | 1

BASELINE CHARACTERISTICS:
Population: Revision patients treated with NuVent
Arm/Group | NuVent™
Number analyzed (Participants) | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.6 (14.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 50
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 44
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 51

OUTCOME MEASURES:

1. Primary Outcome: Navigation to the Desired Sinus Treatment Location and Dilation of the Ostium
Description: Two-fold endpoint: Investigator-assessment regarding the number of sinuses that were easily navigated to the desired treatment location and easy dilation of the ostium
Time Frame: At time of surgery
Population: All patients that completed the study
Measure: Number; unit: Number of sinuses
Arm/Group | NuVent™
Number analyzed (Participants) | 48
Number of sinuses | 121

2. Primary Outcome: Device-related Adverse Event Point Estimate
Description: The primary safety endpoint was the point estimate (and confidence interval) for all AEs that were directly attributable to the device or for which the cause could not be determined and that met the definition of designated primary safety endpoint AEs as defined in the protocol.
Time Frame: 2 weeks
Population: Participants
Measure: Number (95% Confidence Interval); unit: Adverse Events
Arm/Group | NuVent™
Number analyzed (Participants) | 51
Adverse Events | 0 [0 to 3.00]

3. Secondary Outcome: Device Safety Profile as Measured by the Overall Adverse Event Rate
Description: Overall adverse event rate
Time Frame: 2 weeks
Measure: Number; unit: Percentage of participants with an AE
Arm/Group | NuVent™
Number analyzed (Participants) | 51
Percentage of participants with an AE | 18

ADVERSE EVENTS:
Arm/Group | NuVent™
Serious Adverse Events (participants affected / at risk) | 0/51
Other Adverse Events (participants affected / at risk) | 0/51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days